CLINICAL TRIAL: NCT01475656
Title: Safety, Tolerability, and Efficacy of Levetiracetam for Neonatal Seizures
Brief Title: Efficacy of Keppra for Neonatal Seizures
Status: Terminated | Type: Observational
Why Stopped: difficulty with recruitment
Sponsor: Stephanie Merhar, MD (Other)
Responsible Party: Sponsor-Investigator, Stephanie Merhar, MD, Assistant Professor of Pediatrics, Children's Hospital Medical Center, Cincinnati
Organization: Children's Hospital Medical Center, Cincinnati (Other)
Other Study IDs: 2011-1557
Record Dates: First submitted 2011-11-17; First posted 2011-11-21 (Estimated); Last update posted 2013-04-19 (Estimated); Status verified 2013-04

CONDITIONS: Neonatal Seizures
MeSH Terms: interventions — Levetiracetam

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Levetiracetam as first line: Babies who receive levetiracetam as a first line drug for seizures
  Interventions: Drug: levetiracetam
- Phenobarbital as first line: Babies who receive phenobarbital as a first line drug for seizures and levetiracetam as a second line drug
  Interventions: Drug: levetiracetam

INTERVENTIONS:
Drug: levetiracetam — Infants in the both groups will receive 50 mg/kg IV levetiracetam after (continued) seizures are EEG confirmed.

SUMMARY:
The purpose of this research study is to learn how well the medication levetiracetam (Keppra) works to treat seizures in full term and premature babies. Levetiracetam is commonly used in babies with seizures at Cincinnati Children's Hospital, especially if the seizures have not been stopped by other medicines. The Food and Drug Administration (FDA) has approved the use of levetiracetam for older children (over the age of 4) but not for infants. Even though it is not FDA approved for this age group, doctors at Cincinnati Children's use the medicine as a second drug in babies whose seizures are not stopped by phenobarbital. Some doctors are concerned that phenobarbital is not the best medicine to treat seizures in babies, so researchers are trying to study other medicines.

In this study, the investigators are looking at how well levetiracetam stops or slows down seizures in babies. The investigators are also studying the blood levels of levetiracetam to learn more about how the medicine is processed by the body and what level of medicine in the body works to stop seizures. The investigators are checking labs before and after giving the dose to make sure the medication does not cause any changes in blood counts, kidney function, or liver function. The investigators are following all of the babies in the study after hospital discharge to see if the parents notice any side effects of the medication. Babies in the study will come back to the High Risk Follow Up Clinic at Cincinnati Children's at 6 months of age for a visit with a neurologist and a neonatologist and developmental testing.

ELIGIBILITY:
Inclusion criteria:

* Gestational age ≥ 35 weeks
* Postnatal age ≤ 30 days
* Birth weight ≥ 2000 grams
* Clinical or electrographic seizures of any etiology requiring treatment with an antiepileptic medication (as per the judgment of the clinician caring for the patient)
* Parental consent obtained

Exclusion criteria:

* Infants with renal insufficiency indicated by serum creatinine > 2.0 (as part of pre-screening, labs obtained as part of routine care will be reviewed. Infants who have not had a creatinine drawn will have one drawn as part of the study after consent is obtained. If the baby requires levetiracetam emergently before the results of the creatinine are back, the dose will still be given and levels will still be drawn as per the protocol.
* Infants who have previously received levetiracetam
* Parents refuse consent

Max Age: 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 25 neonates ≥ 35 weeks of gestation and ≤ 30 days of life with electrographically-confirmed seizures
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2011-11; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Efficacy | 24 hours
  The primary outcome is the proportion of infants who achieve electrographic seizure freedom as measured by continuous EEG monitoring for 24 hours after intravenous levetiracetam administration.

SECONDARY OUTCOMES:
Pharmacokinetics | 24 hours
  Pharmacokinetic parameters and the concentration-response relationship will be determined by collecting 3 blood samples in the 24 hours after the dose (2-15 minutes post infusion, 1-2 hours post infusion, and 6-10 hours post infusion).
Safety | 7 days
  Safety will be monitored by reviewing changes in vital signs and laboratory parameters after the dose.
Tolerability | 6 months
  Infants who remain on levetiracetam after discharge will be followed for 6 months to determine post-hospital treatment-emergent adverse events. All infants in the study will receive a 6 month developmental profile using the Bayley Scales of Infant Development.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie L Merhar, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States